CLINICAL TRIAL: NCT07297095
Title: The Effect of Virtual Reality Education on Preoperative Anxiety, Postoperative Pain, and Sleep in Patients Undergoing Colon Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08/832
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Preoperative Anxiety; Virtual Reality; Postoperative Pain Management; Postoperative Sleep
Keywords: virtual reality; preoperative anxiety; postoperative sleep; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Participants in the intervention group will receive training in the patient room of the General Surgery Clinic using a training video prepared with virtual reality glasses. The training video will include an introduction to the devices used in the ward during the preoperative period, from blood pressure cuffs to monitors. On the first postoperative day, the Richards Campbell Sleep Scale will be administered to the intervention and control groups. At 8, 16, and 24 hours, the intervention and control groups will be assessed for pain intensity using the Visual Analog Scale (VAS).
  Interventions: Other: preoperative patient education via virtual reality device
- control group (No Intervention): The control group will receive routine verbal training as applied in the classical hospital procedure. The control group will receive routine verbal training as applied in the classical hospital procedure.

INTERVENTIONS:
Other: preoperative patient education via virtual reality device — In the General Surgery Clinic, intervention group participants will receive training in the patient room using a virtual reality headset. The training video will include an introduction to the devices used in the ward during the preoperative period, from blood pressure cuffs to monitors. A training video will be prepared explaining that the patient will be monitored upon returning to the room after the surgery, will be monitored frequently, will be questioned about pain and sleep, and that their family and nurse will be available for any needs they may have.
  Arms: experimental

SUMMARY:
The effect of patient education given to patients undergoing colon surgery using virtual reality in the preoperative period on preoperative anxiety, postoperative pain and sleep is the subject of this study.

DETAILED DESCRIPTION:
This study will be conducted to investigate the effects of patient education provided through virtual reality in the preoperative period to patients undergoing colon surgery on preoperative anxiety, postoperative pain, and sleep. The population of this randomized controlled experimental study will consist of patients who will undergo colon surgery in the General Surgery Department of a university hospital after obtaining ethics committee and institutional approval. The population of the study will consist of patients who will undergo colon surgery in the General Surgery Department of a university hospital after obtaining ethics committee and institutional approval. The required sample size and power calculations for this study were made using the G*Power 3.1.9.2 program. A type 1 error of 0.05, a confidence interval of 90%, and an effect size of 0.72 (Uğraş et al., 2023) were calculated. In the calculation, 41 patients were calculated for each of the intervention and control groups, and the number was increased by 10% to account for losses, with 45 patients each, for a total of 90 patients. "Patient Information Form", "Surgical Anxiety Scale", "Richard Campbell Sleep Scale", "Visual Analog Scale (VAS)" will be used as data collection tools. After completing the "Patient Information Form" on patients who provided informed consent, the "Surgical Anxiety Scale" will be administered to patients in the intervention and control groups upon admission. The intervention group will receive training using a 3D animated patient education video prepared with virtual reality glasses. The control group will receive routine verbal education. Following the training, the "Surgical Anxiety Scale" will be administered a second time to patients. Postoperative pain and sleep assessments will then be conducted in both the control and intervention groups. Pain intensity will be measured with the Visual Analog Scale (VAS) at the 8th, 16th, and 24th postoperative hours for both groups. Postoperative sleep quality will be assessed with the "Richard Campbell Sleep Scale" at the 24th postoperative hour for both groups. IBM SPSS Statistics 22.0 will be used for data analysis and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study will be included:

They are undergoing surgery for the first time,

They have not received preoperative training,

They will undergo colon surgery,

They are over 18 years of age,

They are eligible for the Virtual Reality Discomfort Questionnaire,

They do not have claustrophobia.

Exclusion Criteria:

* Patients who have had multiple surgeries, Patients with head and neck, vision, or hearing problems that prevent them from wearing virtual reality glasses, Patients who had a stoma created during surgery, Patients who wish to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) Richard Campbell Sleep Quality Scale Surgical Anxiety Scale | 6 month
  The Visual Analog Scale (VAS) will be used in the study to assess patients' pain. It is a simple, effective, repeatable, and minimally instrumental measurement tool.
  Richard Campbell Sleep Quality Scale Developed by Richards, this six-item scale measures the depth and quality of nighttime sleep, time to fall asleep, frequency of awakenings and duration of wakefulness, and ambient noise.
  Surgical Anxiety Scale The scale has three subscales: health-related anxiety, recovery-related anxiety, and procedure-related anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Koçaşlı, Assist. Prof. Dr., Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No